CLINICAL TRIAL: NCT03676101
Title: A Randomized, Double-Blind and Placebo-Controlled Phase I Study to Evaluate the Safety and Primary Immunogenicity of the 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha) in Chinese Female Subjects Aged 9-45 Years
Brief Title: Evaluate the Safety and Primary Immunogenicity of 9-valent HPV Recombinant Vaccine in Chinese Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Collaborators: Chongqing Bovax Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9-HPV-1001
Record Dates: First submitted 2018-09-12; First posted 2018-09-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Cervical Cancers; Vulvar Cancer; Vaginal Cancer; CIN1; CIN2; CIN 3; AIS; Invasive Carcinoma; Mild Dysplasia of Vulva; Moderate Dysplasia of Vulva; Vin III; VaIN1; VaIN2; VaIN3; Genital Wart
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9-valent HPV Recombinant Vaccine (Experimental)
  Interventions: Biological: 9-valent HPV Recombinant Vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 9-valent HPV Recombinant Vaccine — Subjects received 3 doses of 9-valent HPV vaccine according to a 0, 2, 6-month schedule.
  Arms: 9-valent HPV Recombinant Vaccine
Biological: Placebo — Subjects received 3 doses of Placebo according to a 0, 2, 6-month schedule.
  Arms: Placebo

SUMMARY:
To evaluate the safety and immunogenicity of the 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha) in Chinese Female Subjects Aged 9-45 Years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females between, and including, 9 and 45 years of age at the time of enrolment
* Be able to provide legal identification for the sake of recruitment
* Be able to understand and sign informed consent form prior to enrollment and for subjects aged 9-17 years, they and their legal guardian(s) are supposed to understand and sign informed consent form together
* Subjects who the investigator believes that they can and will comply with the protocol requirements
* Subject must be not pregnant at the enrollment and agree to use adequate contraceptive precautions within 7 months or don't have pregnancy plan

Exclusion Criteria:

* Fever or axillary temperature> 37.0℃ before vaccination
* Previous vaccination against HPV
* Planned administration/administration of investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding first dose of vaccine
* Planned to take part in other clinical research within 7 months after participating this study or have taken part in other clinical research within 3 months before participating this study
* Abnormal laboratory tests parameters(except the part the clinician diagnosed as non clinical significance)
* Administration of any whole blood, plasma or immunoglobulins products within 3 months preceding first vaccination
* Interval between administration of the study vaccination and any attenuated live vaccine less than 14 days, and other vaccines less than 10 days
* History of serious allergic disease requiring medical intervention (such as oral and throat swelling, difficulty breathing, hypotension or shock)
* History of to adverse event to vaccine, or allergic to some food or drug
* History of epilepsy, seizures or convulsions, or family history of mental illness
* Subjects are immunocompromised or have been diagnosed as suffering from congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis inflammation (JRA), inflammatory bowel disease or other autoimmune diseases, administration of immunosuppressants with six months prior to the first vaccine dose.
* Asplenia, functional asplenia, or any circumstances result of asplenia or splenectomy
* Subject to severe hepatorenal disease, cardiovascular disease, hypertension, diabetes, malignant tumor, all kinds of infectious diseases and acute illness, or during chronic disease acute attack period
* Medical diagnosis of coagulation abnormalities (eg, clotting factor deficiency, coagulation disorders, platelet anomaly) or obvious bruising or coagulation disorder
* Breastfeeding, pregnancy (including pregnancy test positive), or planned to be pregnant within 7 months
* During acute disease (including infectious and non-infectious disease) and chronic diease period of onset
* Abnormal cervical cancer screening or subject to CIN or acuteness wet wart that relevant to HPV infection in the past two years
* Planned to move out of local before the end of the study or leave the local for a long time during the study period
* Other unsuitable factors for the study judged by investigators

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Number of Subjects Reporting Solicited Adverse Events | 7 days after each vaccination
Number of Subjects Reporting Unsolicited Adverse Events | 30 days after each vaccination
Number of Subjects Reporting Serious Adverse Events | 30 days after third dose of vaccination

SECONDARY OUTCOMES:
Geometric Mean Titers (GMTs) to HPV Types 6/11/16/18/31/33/45/52/58 | 30 days after third dose of vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial Center for Disease Control and Prevention, Hanzhou, China